CLINICAL TRIAL: NCT02581826
Title: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Brief Title: Safety and Efficacy of Silodosin in the Treatment of Premature Ejaculation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Cheng-Hsing Hsieh, Cheng-Hsing Hsieh, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-X15-058
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silodosin (Active Comparator): 1. Silodosin capsules of 4 mg, oral: 4 mg once daily with a meal, total dosage 12 mg for 14-21 days.
  2. This arm received Silodosin in the first intervention period and Placebo in the second period (after washout period of 14-21 days).
  3. The patients received 4 mg of Silodosin 1 times a day, total dosage 12 mg for 14-21 days.
  Interventions: Drug: Silodosin
- Placebo (Placebo Comparator): 1. Placebo capsules of 4 mg, oral: 4 mg once daily with a meal, total dosage 12 mg for 14-21 days.
  2. This arm received Placebo in the first period and Silodosin in the second period (after washout period of 14-21 days).
  3. The patients received 4 mg of Placebo 1 times a day, total dosage 12 mg for 14-21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin — α1-adrenoceptor antagonists are distributed not only in the bladder neck, urethra, and prostate, but also in the seminal vesicle and vas deferens. Specifically, the distribution of messenger ribonucleic acid (mRNA) of α1-adrenoceptor antagonists in seminal vesicle and vas deferens is reported to be 75-97%. It is reasonable to use α1-adrenoceptor antagonists with high selectivity for patients with Premature Ejaculation (PE). A new highly selective α1-adrenoceptor antagonists, is strongly associated with dry ejaculation with loss of seminal emission. It had the highest selectivity for the vas deferens compared with other α1-adrenoceptor antagonists.The effectiveness of highly selective α1-adrenoceptor antagonists as a potential therapy for this class of patients was scarcely investigated.
  Other Names: Urief
  Arms: Silodosin
Drug: Placebo — No column specified.
  Arms: Placebo

SUMMARY:
The objectives of the present study aims to evaluate the safety and efficacy of Silodosin in a population of patients wih Premature Ejaculation (PE). Coupled with efficient diagnosis, it is hoped that the newer agent will improve the quality of life for patients who suffer from Premature Ejaculation (PE).

DETAILED DESCRIPTION:
Premature Ejaculation (PE) is characterized as the most common sexual dysfunction in men with a prevalence of 21-33%. Based on the main theories about the pathophysiology of Premature Ejaculation (PE), the most commonly prescribed medications are topical anesthetics and serotonin-specific reuptake inhibitors (SSRIs). It has been reported that the abnormal ejaculation of semen is a typical but rather infrequent side effect of some α1-adrenoceptor antagonists. Silodosin had the highest selectivity for the vas deferens compared with other α1-adrenoceptor antagonists.

Patients suitable for inclusion in the baseline period were those who (as part of the Premature Ejaculation Diagnostic Tool (PEDT) questionnaire) rated their perceived control over ejaculation as 'moderately difficult', 'very difficult' or 'extremely difficult', and the other four items as 'about half the time', 'more than half the time' or 'almost always or always'. Patients completed the Index of Premature Ejaculation (IPE) and Premature Ejaculation Profile (PEP) questionnaires, and rated the quality of their orgasm in response to the question: 'In general, how do you rate the orgasm you experience during sexual intercourse?' on a 5-point scale ('very poor', 'poor', 'satisfactory', 'good', 'very good'). Patients with a baseline Intravaginal Ejaculation Latency Time (IELT) of 2 minutes or less, as measured by a partner-held stopwatch, for at least two of the first three sexual encounters were eligible for randomization into the double-blind phase. In total of 40 eligible patients were randomized to receive double-blind treatment with 4 mg Silodosin or matched placebo for 3 months. One dose was to be taken 2 hours before anticipated sexual intercourse, and only one dose was allowed per 24-h period. Ejaculation-delaying techniques and behavioural therapy were to be avoided. Couples were instructed to attempt sexual intercourse four or more times per month during the 12-week treatment period (minimum of 24 h between doses of medication). During each sexual encounter, the Intravaginal Ejaculation Latency Time (IELT) was measured and recorded, together with efficacy and tolerability data. Ejaculation occurring before penetration was assigned an Intravaginal Ejaculation Latency Time (IELT) of 0 minute. The time noted on the stopwatch at this point was recorded as the duration of sexual intercourse until ejaculation or withdrawal. Patients returned to the clinic at 14-21 days intervals (visits 1, 2, 3, 4, 5 and 6) at which the Index of Premature Ejaculation (IPE) and Premature Ejaculation Profile (PEP) questionnaires were completed. Also, at visit 3 and 6 patients had a safety evaluation and rated the quality of their orgasms. Patients' satisfaction for the treatment was evaluated by Clinical Global Impression of Change (CGIC) in Premature Ejaculation (PE).

ELIGIBILITY:
Inclusion Criteria:

* Premature Ejaculation (PE) diagnosed by Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM-IV-TR) criteria.
* Stable heterosexual, monogamous relationships more than 3 months.
* Age of 20 years or order.
* Written informed consent.

Exclusion Criteria:

* α1-adrenoceptor antagonists within 4 weeks.
* Erectile dysfunction (ED) defined by an Index of Erectile Function (IIEF-5) score < 21.
* History of physical or psychological disorder (patient or partner).
* Patient need to adjust dosage during the screening and treatment period, including tricyclic antidepressants, monoamine oxidase inhibitors or selective serotonin reuptake inhibitors (SSRIs).
* Antidepressant therapy, local anaesthetic spray, intracavernosal injection or psychotherapy within 4 weeks.
* History of alcohol or drug abuse.
* Pregnant partners.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Intravaginal Ejaculatory Latency Time (IELT) | up to 12 weeks

SECONDARY OUTCOMES:
Erectile function domain of the International Index of Erectile Function (IIEF) | Baseline
Premature Ejaculation Diagnostic Tool (PEDT) | Baseline
Index of Premature Ejaculation (IPE) | up to 12 weeks
Premature Ejaculation Profile (PEP) | up to 12 weeks
Clinical Global Impression of Change (CGIC) | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsing Hsieh, MD, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Cheng-Hsing Hsieh, Taipei, Xindian, Taiwan